CLINICAL TRIAL: NCT02659046
Title: The Effect of Different Emergency Medical Systems on the Prognosis of Traumatic Brain Injury
Brief Title: Prehospital Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R15158
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FH30: Patients treated by Pirkanmaa physician-staffed emergency medical service (EMS) unit
- FH10: Patients treated by Helsinki and Uusimaa physician-staffed emergency medical service (EMS) unit

SUMMARY:
The aim of the study is to measure the effect of Finnish physician-staffed EMS unit treatment methods on traumatic brain injury (TBI) patient prognosis.

In the second part of the study the gathered data will be combined with the data from an earlier study (NCT01454648) for regression analysis. The aim of the second study is to identify prehospital factors influencing the prognosis of prehospital TBI patients.

DETAILED DESCRIPTION:
A secondary aim is to identify out-of-hospital treatment factors that can be influenced by education and protocols.

ELIGIBILITY:
Inclusion Criteria:

* TBI with GCS ≤ 8 or unconsciousness verified by an on-call neurosurgeon during admission to the hospital

Exclusion Criteria:

* Multiple trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year

SECONDARY OUTCOMES:
Glasgow outcome score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, Professor, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pakkanen T, Kamarainen A, Huhtala H, Silfvast T, Nurmi J, Virkkunen I, Yli-Hankala A. Physician-staffed helicopter emergency medical service has a beneficial impact on the incidence of prehospital hypoxia and secured airways on patients with severe traumatic brain injury. Scand J Trauma Resusc Emerg Med. 2017 Sep 15;25(1):94. doi: 10.1186/s13049-017-0438-1. PMID 28915898